CLINICAL TRIAL: NCT04456582
Title: Noninvasive Assessment of Myocardial Stiffness by 2D-SWE Ultrasound Technique (Bidimensional Shear Wave Elastography) in Patients With Transthyretin Amyloidosis
Acronym: ELAST-2D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fábio Fernandes (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Fábio Fernandes, Full Professor, University of Sao Paulo General Hospital
Organization: University of Sao Paulo General Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 4963/19/182
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Amyloidosis
Keywords: Amyloidosis; Elastography; Cardiac; Miocardical stiffness
MeSH Terms: conditions — Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Amyloidosis transthyretin with cardiac commitment (Experimental): Shear wave elastography (SWE) will be used to evaluate to assess miocardial elasticity.
  Interventions: Procedure: Shear wave elastography
- Amyloidosis transthyretin without cardiac commitment (Experimental): Shear wave elastography (SWE) will be used to evaluate to assess miocardial elasticity.
  Interventions: Procedure: Shear wave elastography
- Healthy subjects (Placebo Comparator): Shear wave elastography (SWE) will be used to evaluate to assess miocardial elasticity.
  Interventions: Procedure: Shear wave elastography

INTERVENTIONS:
Procedure: Shear wave elastography — The elastographic technique by ultrasound (USE), shear waves or shear wave elastography (SWE), quantitatively evaluates tissue stiffness by mapping the propagation of acoustic waves (shear waves), in a non-invasive manner and without emission of ionizing radiation. Their speeds are tracked by the ultrasound equipment after tissue deformation occurs, generated by pulses of acoustic radiation (ARFI) of the transducer itself. Assuming the correlation between tissue stiffness and increased acoustic propagation speeds, it is possible to describe mathematically the elasticity of tissues by measuring specific acoustic waves.

SUMMARY:
Amyloidosis by mutation of the transthyretin gene (ATTRh) is part of a group of diseases in which the deposit of structurally abnormal proteins (amyloid fibrils) affects multiple organs such as: liver, kidney, eyes, nervous system, gastrointestinal tract and heart, and, finally, it increases the morbidity and mortality of affected patients. This deposit in the myocardium is manifested syndromically as heart failure with preserved or slightly reduced systolic function, and important diastolic dysfunction. The analysis of diastolic function comprises two components: the assessment of active relaxation, dependent on preload and afterload, and the assessment of the passive properties of the tissue - its hardness or rigidity. Myocardial stiffness represents an important parameter for diagnosis and prognosis, but its evaluation is not included in conventional echocardiography. Cardiac elastography has recently been proposed as a non-invasive diagnostic modality to assess myocardial stiffness.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of HRTR with and without cardiac involvement.
* For the definition of cardiac involvement by ATTRh, all the criteria below must be presented:

  * Pathogenic mutation of TTR consistent with ATTRh.
  * Evidence of cardiac commitment by echocardiography or nuclear magnetic resonance with measurement of the interventricular septum at the end of diastole (SIVd)> 12mm or / and medical history of heart failure, and / or levels of troponin and / or BNP above the reference value without another more likely cause.
  * Amyloid deposit in cardiac or extra-cardiac tissue (eg, abdominal fat aspirate, salivary gland, connective sheath of the median nerve) confirmed by congo red staining or presence of grade 2 or 3 myocardial scintigraphy (DPD-CT) of cardiac uptake, in cases where the presence of monoclonal gammopathy of undetermined significance (MGUS) was ruled out.
  * In the presence of MGUS, confirmation of the TTR protein in the tissue is necessary through immunohistochemistry (IHC) or mass spectrometry.

Exclusion Criteria:

* Presence of another type of cardiomyopathy such as hypertension, valve or ischemic heart disease (eg, previous myocardial infarction documented with myocardial necrosis markers and electrocardiographic changes).
* Presence of diseases other than cardiac amyloidosis, impairing the assessment of functional capacity, such as chronic obstructive pulmonary disease, severe arthritis or peripheral arterial disease, recent or planned orthopedic procedure during the course of the study (eg, spine surgery or under lower limbs) that impairs walking in the 6-minute test evaluation.
* Acute coronary heart disease or unstable angina in the past 3 months
* Report of disease of the sinus or atrioventricular node with indication of a pacemaker, but with no intention of implantation.
* Presence of untreated hypothyroidism or hyperthyroidism.
* Previous heart, liver or other organ transplant.
* Presence of neoplasia in the last 3 years, except for basal and squamous cell carcinomas of skin or cervical cancer in situ previously treated.
* Presence of other medical conditions or comorbidities that, in the investigator's opinion, could interfere with the course of the study or the interpretation of the data.
* Pregnancy.
* History of alcohol abuse in the last 2 years or excessive daily alcohol intake (for women, more than 14 units per week; for men, more than 21 units of alcohol per week [unit: one glass of wine (125ml) = one dose of distillate = 332.5ml of beer).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-03 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-05-29 (Estimated)

PRIMARY OUTCOMES:
Dyastolic miocardical elasticity | Around 6 months
  Diastolic myocardial elasticity could provide a more direct response to the constitution of the tissue and allow a simple, safe and diastolic function assessment and early initiation of specific treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo Medical School - The Heart Institute, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No